CLINICAL TRIAL: NCT01022528
Title: Analgesic Effect of Preoperative Dexamethasone in Gynecological Laparotomies - a Dose-ranging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-0005-B
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Fatigue
Keywords: Elective total abdominal hysterectomy (with or without salpingo-oophorectomy or minor bladder repair) or myomectomy; through a lower transverse or low midline incision under general anesthesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Fatigue | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone (0.1 mg/kg); Drug: Dexamethasone (0.2 mg/kg)
- Saline (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Dexamethasone (0.1 mg/kg)
  Other Names: Dose = 0.1 mg/kg
  Arms: Dexamethasone
Drug: Dexamethasone (0.2 mg/kg)
  Other Names: Dose = 0.2 mg/kg
  Arms: Dexamethasone
Other: Saline
  Arms: Saline

SUMMARY:
The objective of the study is to examine the effect of the addition of intravenous dexamethasone 1.5 hours prior to induction of anesthesia on the post-operative opioid consumption, pain scores, fatigue, and recovery in patients undergoing gynecological surgery with laparotomy under general anesthesia.

This is a dose finding study with two different doses (0.1 mg/kg vs. 0.2 mg/kg) of dexamethasone to find out the optimal efficacious dose of dexamethasone with minimal side effects.

Dexamethasone has anti-inflammatory, immunomodulatory, and analgesic effects; and is superior to placebo in providing post-operative pain control, lower analgesic consumption, prevention of postoperative nausea and vomiting, lesser post-operative fatigue, and better recovery profile. No dose response study has been done. The investigators hypothesize that a higher dose of dexamethasone may have an incremental beneficial effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be non-lactating
* 18-65 years of age
* ASA groups I-III for elective total abdominal hysterectomy (with or without salpingo-oophorectomy or minor bladder repair)or myomectomy through a lower transverse or low midline incision under general anesthesia. Incidental appendectomy and /or abdominal lipectomy were allowed as collateral surgical procedures if the same incision was used

Exclusion Criteria:

* Emergent procedures
* Diagnosed malignancy
* History of allergy to dexamethasone
* Allergy or contraindication to drugs used in study and anesthesia
* Patients with uncontrolled diabetes mellitus, recent history of gastrointestinal bleeding or ulceration within 30 days before the study)
* Patients who have taken drugs in the 12 hours preceding the surgery that could confound the analgesic response (specifically analgesics, neuroleptics, corticosteroids, NSAIDs)
* Patients who have been on long term oral steroid therapy
* Patients with BMI>40
* Serious organ disease/ dysfunction
* Chronic pain patients requiring >30mg morphine per day or equivalent
* Severe psychiatric disease
* Drug Addiction
* Pregnancy
* Language barrier
* Inability to cooperate with the use of the intravenous PCA morphine pump

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Total cumulative morphine consumption via the patient-controlled analgesia (PCA) pump in the first 24 hours

SECONDARY OUTCOMES:
Total cumulative postoperative morphine consumption after 48 hours
Numerical Rating Scale at rest (supine) and on movement (on sitting) at baseline, 1, 6, 12, 24 and 48 hours after surgery
Total fentanyl administration intraoperatively and in the PACU
Time to first analgesic request in the PACU
Time to discharge from the PACU

CONTACTS AND LOCATIONS:
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada